CLINICAL TRIAL: NCT03316157
Title: Exercise and Nutritional Rehabilitation in Patients With Cancer, Randomised (1:1) Unblinded Feasibility Trial of a Rehabilitation Programme (Exercise and Nutrition) Versus Waiting List Control, in Patients With Advanced Cancer
Brief Title: Exercise and Nutritional Rehabilitation in Patients With Cancer
Acronym: ENeRgy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Marie Curie Hospice, Belfast (Other); Accord Clinical Research (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AC17085
Record Dates: First submitted 2017-09-22; First posted 2017-10-20 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Cachexia; Cancer; Diet Modification; Physical Activity; Advanced Cancer
MeSH Terms: conditions — Cachexia; Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised (1:1) unblinded feasibility trial of a rehabilitation programme (exercise and nutrition) versus waiting list control, in patients with advanced cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation (Experimental): Advanced cancer patients will receive an 8 week rehabilitation intervention consisting of physical exercise and nutritional supplementation, along with standard care
  Interventions: Dietary Supplement: ProSure; Behavioral: Physical Exercise
- Waiting list Control (No Intervention): Standard care alone for the 8 week trial period, followed by participants being offered the rehabilitation programme

INTERVENTIONS:
Dietary Supplement: ProSure — Patients will take 2x 220mL nutritional supplements per day for 8 weeks and be given dietary advice to optimise their nutrition
  Arms: Rehabilitation
Behavioral: Physical Exercise — Patients will receive an individualised exercise regimen consisting of 60 minutes aerobic and 3x resistance elements per week
  Arms: Rehabilitation

SUMMARY:
In patients with incurable cancer, general deterioration in their ability to walk, exercise and care for themselves is often regarded as an inevitable consequence of this. In 2015, Hospice UK published a report advocating "Rehabilitative Palliative Care".

However there is limited robust evidence on which to base this approach. Reviews of the literature show limited study numbers but do suggest that rehabilitation may be feasible for advanced cancer patients. However key components were not clear and no recommendations could be given.

This trial is designed primarily to test the feasibility of a rehabilitation programme (exercise and nutritional supplementation) in advanced cancer patients. Feasibility will be the primary outcome measure including rates of recruitment and compliance. Secondary outcome measures include impact on physical function, nutritional status, quality of life for patients and their carers. We will also assess the health economic impact by assessing patient health facility use throughout the trial.

40 patients with advanced cancer living in the community will be recruited from two hospice palliative care teams in Edinburgh. These patients will be randomised in to either the treatment arm: the rehabilitation programme plus standard care, or the control arm: standard care alone. The treatment arm will consist of an 8 week rehabilitation programme, supervised at weekly clinics by a physiotherapist and dietician.

To minimise contamination the control group will be offered the treatment at the end of the 8 weeks (waiting list control).

Measurements will be made for both groups and compared at baseline (week 0), midpoint (week 5) and endpoint (week 9). Recommendations for a larger UK wide trial will be made from the findings of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced cancer (defined as metastatic or locally advanced cancer not amenable to curative treatment).
2. Outpatient
3. ≥18years
4. Karnofsky score ≥ 60
5. Prognosis greater than 3 months
6. Able to complete trial based assessments
7. Under care of community services at Marie Curie or St Columba's Hospices
8. Ability to comply with trial protocol
9. Ability to provide and have capacity to consent
10. Agree to attend trial centre for trial related activity (St Columba's Hospice)

Exclusion Criteria:

1. Undergoing anti-cancer therapy (hormonal treatment or bisphosphonates permitted)
2. Using enteral nutrition (NG or similar) or parenteral nutrition
3. Co-enrolment in drug trials
4. Inability to swallow

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of Rehabilitation programme | 8 weeks
  Compliance with treatment and trial procedures

SECONDARY OUTCOMES:
Patient quality of life | 8 weeks
  Measured by EORTC QLQ-C15-PAL questionnaire
Carer quality of life | 8 weeks
  Measured by CQOLC questionnaire
Change in physical function | 8 weeks
  Mean daily step count, measured by Physical Activity Meter over 5 days
Change in physical function | 8 weeks
  Measured by two-minute walk test (metres/feet covered)
Change in physical function | 8 weeks
  Measured by Karnofsky performance status (KPS) at baseline, mid and endpoint
Change in physical function | 8 weeks
  Measured by timed up-and-go test (Seconds)
Change in physical function | 8 weeks
  Measured by Life Space Assessment scores
Sleep quality | 8 weeks
  Measured by physical activity meter at baseline and endpoint (Mean sleep hours, mean hours restless and hours awake)
Nutritional status | 8 weeks
  Height and weight measured at baseline, mid and endpoint assessment (m, Kg and combined as kg/m2)
Nutritional status | 8 weeks
  Measured by PG-SGA nutritional assessment (PG-SGA point score)
Contamination in the control group | 8 weeks
  Measured by dietary intake using 24 hour recall (patient diary entries)
Contamination in the control group | 8 weeks
  Measured by change in measures of physical function (see outcomes 4-8) in control group from baseline measurement to endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom